CLINICAL TRIAL: NCT00892983
Title: Primary Prevention of Rapid Weight Gain in Early Childhood: a Randomised Controlled Trial
Brief Title: Prevention of Overweight in Infancy
Acronym: POInz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: Health Research Council of NZ (Unknown)
Responsible Party: Principal Investigator, Barry Taylor, Professor, University of Otago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 105891.01.P.NH; HRC 08/374 (Other Grant/Funding Number: NZ Health Research Council)
Record Dates: First submitted 2009-05-03; First posted 2009-05-05 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Growth; Sleep
Keywords: Obesity; Sleep; Physical activity; Breast feeding; Depression
MeSH Terms: conditions — Obesity; Motor Activity; Breast Feeding; Depression | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard well child care (No Intervention): Standard Well Child Care (SWCC) - 8 Core visits at 2-4 weeks, 6 weeks, 3, 5, 8-10 and 15 months, 2 and 3 years.
- Food Activity Breast feeding support (Experimental): FAB (Food Activity Breast feeding support) 8 extra parent contacts for augmented education and support around breast feeding, food and activity
  Interventions: Behavioral: FAB
- Sleep (Experimental): Prevention of sleep problems in first 6 months and then active early intervention for sleep problems from 6 months to 24 months
  Interventions: Behavioral: Sleep
- FAB + Sleep (Experimental): combination of interventions used in arms 2 and 3
  Interventions: Behavioral: FAB; Behavioral: Sleep

INTERVENTIONS:
Behavioral: FAB — Standard well child care plus 7 extra parent contacts for augmented education and support around breast feeding, food and activity with 1 before birth and then at 1-2 weeks, and 3, 4, 7, 9, 13, and 18 months post-partum.
  Arms: FAB + Sleep; Food Activity Breast feeding support
Behavioral: Sleep — Standard well child care plus 2 extra contacts focussed on Sleep with 1 before birth (anticipatory guidance), and sleep problem prevention at 3 weeks. A sleep problem intervention starting at 6 months was possible for those indicating their child had a sleep problem at 6 months of age. Main prevention advice focussed on placing baby to sleep awake, maximising night-day differences and use of sleep place in parents bedroom for first 6 months. Intervention after 6 months uses preferentially a technique called "parental presence", and if this does not fit family a technique called "camping out" and finally, if neither of the first two fit family, controlled crying.
  Arms: FAB + Sleep; Sleep

SUMMARY:
Obesity is one of the biggest threats to health in the 21st century. Rapid weight gain in the first year of life tends to lead to overweight in children, which in turn leads to overweight in adults. This rapid early weight gain occurs most often at weaning when eating patterns emerge. Infant sleep problems also appear to be associated with the risk of becoming overweight, and contribute to maternal post-natal depression. We propose to undertake a 4-arm randomised controlled trial to determine whether extra education and support for families around weaning and development of early food and activity habits, with or without intervention to improve infant sleep, will decrease the current risk patterns of rapid excessive early childhood weight gain in New Zealand. This would provide strong evidence for the value of such a strategy in the long term control of the obesity epidemic and its consequent complications.

This is a two-year intervention with follow-ups at 3.5, 5 and 11 years of age.

DETAILED DESCRIPTION:
We plan on undertaking a 4-arm randomised controlled trial to test the following hypotheses:

1. That anticipatory guidance and extra education and support in infancy around weaning and decreasing/avoiding television watching will delay the timing of introduction of solid foods, will be associated with more successful introduction of nutrient dense foods with appropriate portion size and decrease small screen exposure leading to a lower number of children with excessive weight velocity in infancy and early childhood.
2. That anticipatory guidance, education and extra support around the early development of infant sleeping patterns will decrease sleep problems, increase infant sleeping time, decrease arousals at night and lower sleep latency which will in turn influence rate of early infant weight gain.
3. That interventions 1 and 2 will interact additively with regard to infant and early childhood weight gain.
4. That intervention 2 will lead to lower rates of maternal depression and increased family well being.

ELIGIBILITY:
Inclusion Criteria:

* Mothers booked for delivery in Dunedin, New Zealand

Exclusion Criteria:

* Women booked after 34 weeks gestation,
* Identified congenital abnormality likely to affect feeding and/or growth
* Home address outside of metropolitan Dunedin or Invercargill,
* Families who are likely to shift out of metropolitan Dunedin or Invercargill in the next 2 years.
* Unable to communicate in English or te reo Maori.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 802 (Actual)
Dates: Start 2009-05; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
BMI z score | 24 months (end of intervention)
  BMI z score derived from ht and weight and using World Health Organisation (WHO) growth standards
BMI z score | 60 months of age (followup at 5 years of age)
  BMI z score derived from ht and weight and using WHO growth standards
BMI z score | Follow-up at 11 years of age
  BMI z score derived from height and weight and using WHO reference data

SECONDARY OUTCOMES:
Dietary intake | 24 months (end of intervention) and 60 months (end of follow-up) and 11 years (further follow-up)
  Dietary information (foods, food groups, nutrients) via food frequency questionnaire
Television viewing | 24 months (end of intervention) and 60 months (end of follow-up)
  Hours of screen use by parental questionnaire
Major/ Moderate sleep problems | 24 months (end of intervention)
  Parents indicate presence of sleep problems in child
Physical activity (PA) | 24 months (end of intervention) and 60 months (end of follow-up) and 11 years (further follow-up)
  PA measured using actical accelerometry over 5-7 days
Duration of exclusive and any breast feeding | 24 months
  Measured by repeated questionnaire
Parental depression score | Measured at multiple timepoints between pregnancy and 24 months (end of intervention) and 60 months (end of follow-up)
  Edinburgh Postnatal Depression questionnaire
Sleep | 24 months (end of intervention) and 60 months (end of follow-up) and 11 years (further follow-up)
  Measured by questionnaire and accelerometry at multiple timepoints
Number of night awakenings | 24 months (end of intervention) and 60 months (end of follow-up)
  Measured by questionnaire and accelerometry at multiple timepoints
Self-regulation | 42 and 60 months
  Measured by questionnaire and laboratory based measures at follow-up only
Body composition | 60 months and 11 years (further follow-up)
  Measured by dual-energy x-ray absorptiometry at follow-up only

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Taylor, FRACP, Principal Investigator — University of Otago; Rachael Taylor, PhD, Principal Investigator — University of Otago
Locations (1):
- University of Otago, Dunedin, South Island, New Zealand

REFERENCES:
- [Background] Taylor RW, Heath AL, Galland BC, Cameron SL, Lawrence JA, Gray AR, Tannock GW, Lawley B, Healey D, Sayers RM, Hanna M, Meredith-Jones K, Hatch B, Taylor BJ. Three-year follow-up of a randomised controlled trial to reduce excessive weight gain in the first two years of life: protocol for the POI follow-up study. BMC Public Health. 2016 Aug 11;16(1):771. doi: 10.1186/s12889-016-3383-4. PMID 27514714
- [Background] Taylor RW, Iosua E, Heath AM, Gray AR, Taylor BJ, Lawrence JA, Hanna M, Cameron SL, Sayers R, Galland B. Eating frequency in relation to BMI in very young children: a longitudinal analysis. Public Health Nutr. 2017 Jun;20(8):1372-1379. doi: 10.1017/S1368980017000143. Epub 2017 Feb 27. PMID 28238299
- [Background] Galland BC, Sayers RM, Cameron SL, Gray AR, Heath AM, Lawrence JA, Newlands A, Taylor BJ, Taylor RW. Anticipatory guidance to prevent infant sleep problems within a randomised controlled trial: infant, maternal and partner outcomes at 6 months of age. BMJ Open. 2017 Jun 2;7(5):e014908. doi: 10.1136/bmjopen-2016-014908. PMID 28576897
- [Background] Moir C, Meredith-Jones K, Taylor BJ, Gray A, Heath AM, Dale K, Galland B, Lawrence J, Sayers RM, Taylor RW. Early Intervention to Encourage Physical Activity in Infants and Toddlers: A Randomized Controlled Trial. Med Sci Sports Exerc. 2016 Dec;48(12):2446-2453. doi: 10.1249/MSS.0000000000001055. PMID 27471782
- [Background] Fangupo LJ, Heath AL, Williams SM, Somerville MR, Lawrence JA, Gray AR, Taylor BJ, Mills VC, Watson EO, Galland BC, Sayers RM, Hanna MB, Taylor RW. Impact of an early-life intervention on the nutrition behaviors of 2-y-old children: a randomized controlled trial. Am J Clin Nutr. 2015 Sep;102(3):704-12. doi: 10.3945/ajcn.115.111823. Epub 2015 Jul 29. PMID 26224299
- [Background] Cameron SL, Heath AL, Gray AR, Churcher B, Davies RS, Newlands A, Galland BC, Sayers RM, Lawrence JA, Taylor BJ, Taylor RW. Lactation Consultant Support from Late Pregnancy with an Educational Intervention at 4 Months of Age Delays the Introduction of Complementary Foods in a Randomized Controlled Trial. J Nutr. 2015 Jul;145(7):1481-90. doi: 10.3945/jn.114.202689. Epub 2015 May 20. PMID 25995280
- [Background] Meredith-Jones K, Haszard J, Moir C, Heath AL, Lawrence J, Galland B, Taylor B, Gray A, Sayers R, Taylor R. Physical activity and inactivity trajectories associated with body composition in pre-schoolers. Int J Obes (Lond). 2018 Sep;42(9):1621-1630. doi: 10.1038/s41366-018-0058-5. Epub 2018 Mar 15. PMID 29717271
- [Background] Taylor RW, Haszard JJ, Meredith-Jones KA, Galland BC, Heath AM, Lawrence J, Gray AR, Sayers R, Hanna M, Taylor BJ. 24-h movement behaviors from infancy to preschool: cross-sectional and longitudinal relationships with body composition and bone health. Int J Behav Nutr Phys Act. 2018 Nov 26;15(1):118. doi: 10.1186/s12966-018-0753-6. PMID 30477518
- [Background] Taylor RW, Gray AR, Heath AM, Galland BC, Lawrence J, Sayers R, Healey D, Tannock GW, Meredith-Jones KA, Hanna M, Hatch B, Taylor BJ. Sleep, nutrition, and physical activity interventions to prevent obesity in infancy: follow-up of the Prevention of Overweight in Infancy (POI) randomized controlled trial at ages 3.5 and 5 y. Am J Clin Nutr. 2018 Aug 1;108(2):228-236. doi: 10.1093/ajcn/nqy090. PMID 30101329
- [Background] Hatch B, Galland BC, Gray AR, Taylor RW, Sayers R, Lawrence J, Taylor B. Consistent use of bedtime parenting strategies mediates the effects of sleep education on child sleep: secondary findings from an early-life randomized controlled trial. Sleep Health. 2019 Oct;5(5):433-443. doi: 10.1016/j.sleh.2019.03.002. Epub 2019 May 20. PMID 31122876
- [Background] Leong C, Haszard JJ, Heath AM, Tannock GW, Lawley B, Cameron SL, Szymlek-Gay EA, Gray AR, Taylor BJ, Galland BC, Lawrence JA, Otal A, Hughes A, Taylor RW. Using compositional principal component analysis to describe children's gut microbiota in relation to diet and body composition. Am J Clin Nutr. 2020 Jan 1;111(1):70-78. doi: 10.1093/ajcn/nqz270. PMID 31711093
- [Background] Meredith-Jones K, Galland B, Haszard J, Gray A, Sayers R, Hanna M, Taylor B, Taylor R. Do young children consistently meet 24-h sleep and activity guidelines? A longitudinal analysis using actigraphy. Int J Obes (Lond). 2019 Dec;43(12):2555-2564. doi: 10.1038/s41366-019-0432-y. Epub 2019 Sep 2. PMID 31477783
- [Background] Askie LM, Espinoza D, Martin A, Daniels LA, Mihrshahi S, Taylor R, Wen LM, Campbell K, Hesketh KD, Rissel C, Taylor B, Magarey A, Seidler AL, Hunter KE, Baur LA. Interventions commenced by early infancy to prevent childhood obesity-The EPOCH Collaboration: An individual participant data prospective meta-analysis of four randomized controlled trials. Pediatr Obes. 2020 Jun;15(6):e12618. doi: 10.1111/ijpo.12618. Epub 2020 Feb 6. PMID 32026653
- [Background] Roy M, Haszard JJ, Savage JS, Yolton K, Beebe DW, Xu Y, Galland B, Paul IM, Mindell JA, Mihrshahi S, Wen LM, Taylor B, Richards R, Te Morenga L, Taylor RW. Bedtime, body mass index and obesity risk in preschool-aged children. Pediatr Obes. 2020 Sep;15(9):e12650. doi: 10.1111/ijpo.12650. Epub 2020 May 6. PMID 32372572
- [Result] Taylor BJ, Gray AR, Galland BC, Heath AM, Lawrence J, Sayers RM, Cameron S, Hanna M, Dale K, Coppell KJ, Taylor RW. Targeting Sleep, Food, and Activity in Infants for Obesity Prevention: An RCT. Pediatrics. 2017 Mar;139(3):e20162037. doi: 10.1542/peds.2016-2037. PMID 28242860
- [Derived] Taylor RW, Haszard JJ, Meredith-Jones KA, Azeem AA, Galland BC, Heath AM, Taylor BJ, Healey D. Associations between activity, sedentary and sleep behaviours and psychosocial health in young children: a longitudinal compositional time-use study. J Act Sedentary Sleep Behav. 2023 Jan 3;2(1):3. doi: 10.1186/s44167-022-00011-3. PMID 40217436
- [Derived] Taylor RW, Galland BC, Heath AM, Gray AR, Meredith-Jones KA, Fortune SA, Sullivan TA, Adebowale T, McIntosh D, Jackson RF, Taylor BJ. Long-term follow-up of the impact of brief sleep and lifestyle interventions in infancy on BMI z-score at 11 years of age: The POI randomized controlled trial. Pediatr Obes. 2025 Mar;20(3):e13204. doi: 10.1111/ijpo.13204. Epub 2025 Jan 17. PMID 39821586
- [Derived] Taylor RW, Haszard JJ, Healey D, Meredith-Jones KA, Taylor BJ, Galland BC. Adherence to 24-h movement behavior guidelines and psychosocial functioning in young children: a longitudinal analysis. Int J Behav Nutr Phys Act. 2021 Aug 25;18(1):110. doi: 10.1186/s12966-021-01185-w. PMID 34433476
- [Derived] Fangupo LJ, Haszard JJ, Taylor BJ, Gray AR, Lawrence JA, Taylor RW. Ultra-Processed Food Intake and Associations With Demographic Factors in Young New Zealand Children. J Acad Nutr Diet. 2021 Feb;121(2):305-313. doi: 10.1016/j.jand.2020.08.088. Epub 2020 Oct 21. PMID 33500114
- [Derived] Adebowale TO, Taylor BJ, Gray AR, Galland BC, Heath AM, Fortune S, Meredith-Jones KA, Sullivan T, McIntosh D, Brosnan B, Taylor RW. Long-Term Follow-Up of a Randomized Controlled Trial to Reduce Excessive Weight Gain in Infancy: Protocol for the Prevention of Overweight in Infancy (POI) Follow-Up Study at 11 Years. JMIR Res Protoc. 2020 Nov 30;9(11):e24968. doi: 10.2196/24968. PMID 33252344
- [Derived] Haszard JJ, Russell CG, Byrne RA, Taylor RW, Campbell KJ. Early maternal feeding practices: Associations with overweight later in childhood. Appetite. 2019 Jan 1;132:91-96. doi: 10.1016/j.appet.2018.10.008. Epub 2018 Oct 9. PMID 30308224
- [Derived] Taylor BJ, Heath AL, Galland BC, Gray AR, Lawrence JA, Sayers RM, Dale K, Coppell KJ, Taylor RW. Prevention of Overweight in Infancy (POI.nz) study: a randomised controlled trial of sleep, food and activity interventions for preventing overweight from birth. BMC Public Health. 2011 Dec 19;11:942. doi: 10.1186/1471-2458-11-942. PMID 22182309
- See also: University of Otago — http://www.otago.ac.nz